CLINICAL TRIAL: NCT06131125
Title: Comparative Effects of Plyometric and Explosive Strength Training on Agility, Power, and Dynamic Balance in Basketball Players
Brief Title: Plyometric vs Explosive Strength Training on Agility, Power, and Balance in Basketball Players
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR&AHS/23/0439
Record Dates: First submitted 2023-11-09; First posted 2023-11-14 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Plyometric Exercise; Resistance Training; Basketball
Keywords: Plyometric training; Explosive strength training; Basketball
MeSH Terms: interventions — Plyometric Exercise

STUDY DESIGN:
Intervention Model Description: randomized clinical trail
Who Masked: Outcomes Assessor
Masking Description: The assessor who will take the readings is blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plyometric Training (Experimental): Group A will perform plyometric training that includes squats, burpees, box jumps, tuck jumps, skaters hop, single-leg deadlift to jump. 10 reps of 3 sets with three sessions per week for 6 weeks.
  Interventions: Other: Plyometric training exercises
- Explosive Strength Training (Experimental): Group B will perform explosive strength training that includes dumbbell push presses, sprint running, sled pushes, shuttle runs. 10 reps of 3 sets with three sessions per week for 6 weeks.
  Interventions: Other: Explosive strength training exercises

INTERVENTIONS:
Other: Plyometric training exercises — This includes plyometric training exercises thrice a week for 6 weeks
  Arms: Plyometric Training
Other: Explosive strength training exercises — this includes explosive strength training exercises thrice a week for 6 weeks
  Arms: Explosive Strength Training

SUMMARY:
The study is randomized and single-blinded. Ethical approval is taken from Ethical committee of Riphah International University, Lahore. Participants who meet the inclusion criteria will be enrolled and allocated in groups A & B through the sealed envelope method by Non-probability Convenient random sampling technique. Subjects in group A will receive plyometric training. Group B will receive explosive strength training.

DETAILED DESCRIPTION:
The objective of the study is to determine the effects of plyometric training versus explosive strength training on agility, power, and dynamic balance in basketball players. The study is randomized and single-blinded. Ethical approval is taken from the Ethical Committee of Riphah International University, Lahore. Participants who meet the inclusion criteria will be enrolled and allocated in groups A & B through the sealed envelope method by Non-probability Convenient random sampling technique. Subjects in group A will receive plyometric training. Group B will receive explosive strength training. The outcome measures will be assessed by agility T-test, vertical jump test, and star excursion balance test (SEBT).

The data will be analyzed by SPSS, version 25. Statistical significance is p=0.05.

ELIGIBILITY:
Inclusion Criteria:

* Basketball players, both male and female players.
* players aged 17-25 years, players who have been playing basketball for a minimum of two years.

Exclusion Criteria:

* out-of-practice players,
* unwilling participants,
* players with any musculoskeletal injury, and players with any systemic disease.

Ages: 17 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-10-20 (Actual); Primary Completion 2024-02-20 (Estimated); Study Completion 2024-02-20 (Estimated)

PRIMARY OUTCOMES:
agility | pre and 6 weeks post interventional
  agility will be assessed by Agility T-test
power | pre and 6 weeks post interventional
  vertical jump test will be used to measure lower extremity power
dynamic balance | pre and 6 weeks post interventional
  star excursion balance test (SEBT) is used to assess balance

CONTACTS AND LOCATIONS:
Overall Officials: Dawood Emmanuel, DPT, Principal Investigator — Study Principal Investigator
Locations (1):
- City sports Complex, Abbottabad, Khyber Pakhtunkhawa, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mexis D, Nomikos T, Kostopoulos N. Effect of Pre-Season Training on Physiological and Biochemical Indices in Basketball Players-A Systematic Review. Sports (Basel). 2022 May 26;10(6):85. doi: 10.3390/sports10060085. PMID 35736825
- [Background] Santos EJ, Janeira MA. Effects of complex training on explosive strength in adolescent male basketball players. J Strength Cond Res. 2008 May;22(3):903-9. doi: 10.1519/JSC.0b013e31816a59f2. PMID 18438223
- [Background] Matavulj D, Kukolj M, Ugarkovic D, Tihanyi J, Jaric S. Effects of plyometric training on jumping performance in junior basketball players. J Sports Med Phys Fitness. 2001 Jun;41(2):159-64. PMID 11447356
- [Background] Jaksic D, Maricic S, Maksimovic N, Bianco A, Sekulic D, Foretic N, Drid P. Effects of Additional Plyometric Training on the Jump Performance of Elite Male Handball Players: A Systematic Review. Int J Environ Res Public Health. 2023 Jan 30;20(3):2475. doi: 10.3390/ijerph20032475. PMID 36767841
- [Background] Deng N, Soh KG, Huang D, Abdullah B, Luo S, Rattanakoses W. Effects of plyometric training on skill and physical performance in healthy tennis players: A systematic review and meta-analysis. Front Physiol. 2022 Nov 24;13:1024418. doi: 10.3389/fphys.2022.1024418. eCollection 2022. PMID 36505069
- [Background] Ramirez-Campillo R, Garcia-Hermoso A, Moran J, Chaabene H, Negra Y, Scanlan AT. The effects of plyometric jump training on physical fitness attributes in basketball players: A meta-analysis. J Sport Health Sci. 2022 Nov;11(6):656-670. doi: 10.1016/j.jshs.2020.12.005. Epub 2020 Dec 24. PMID 33359798
- [Background] Radenkovic M, Lazic A, Stankovic D, Cvetkovic M, Dordic V, Petrovic M, Tomovic M, Kouidi E, Preljevic A, Markovic J, Beric D, Stojanovic M, Kocic M, Aksovic N, Petkovic E, Coh M, Bogataj S, Bubanj S. Effects of Combined Plyometric and Shooting Training on the Biomechanical Characteristics during the Made Jump Shot in Young Male Basketball Players. Int J Environ Res Public Health. 2022 Dec 26;20(1):343. doi: 10.3390/ijerph20010343. PMID 36612663
- [Background] Santos EJ, Janeira MA. The effects of resistance training on explosive strength indicators in adolescent basketball players. J Strength Cond Res. 2012 Oct;26(10):2641-7. doi: 10.1519/JSC.0b013e31823f8dd4. PMID 22108528
- [Background] King JA, Cipriani DJ. Comparing preseason frontal and sagittal plane plyometric programs on vertical jump height in high-school basketball players. J Strength Cond Res. 2010 Aug;24(8):2109-14. doi: 10.1519/JSC.0b013e3181e347d1. PMID 20634744